CLINICAL TRIAL: NCT04409184
Title: Evaluation of Whole Blood Samples From Coronavirus Disease 2019 (COVID-19) Convalescent Patients to Study Immune Response and Severity of Disease Predictors
Brief Title: Whole Blood Collection From Individuals in the Convalescent Phase of SARS-CoV-2 Infection
Status: Withdrawn | Type: Observational
Why Stopped: Study was not opened.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Versiti Blood Health (Other)
Responsible Party: Principal Investigator, Weiguo Cui, Associate Professor, Microbiology & Immunology, Medical College of Wisconsin
Other Study IDs: PRO00037957
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: COVID; Sars-CoV2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Convalescent subjects: Convalescent, now asymptomatic, subjects with documented prior COVID-19 due to SARS-CoV-2 infection
- Healthy controls

SUMMARY:
The study was not opened.

ELIGIBILITY:
Inclusion Criteria:

Patients who have previously been diagnosed with COVID-19 but are now asymptomatic >14 days and a matched number of healthy controls:

1. Consent: Subject able to provide voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. SARS-CoV-2 Testing Status:

   1. Experimental Population: Subject has had positive SARS-CoV-2 verified by clinical laboratory OR
   2. Control Population: Subject without testing or negative SARS-CoV-2 testing
3. Complete resolution and current absence of clinical symptoms Symptoms Defined as: Fever, Dry cough, Fatigue, Difficulty breathing, Sore throat, Diarrhea, Rhinorrhea (runny nose), or new aches/pains.
4. Age: Greater or equal to 18 years of age. a. Subject must be able to provide voluntary written consent

Exclusion Criteria:

1. Ongoing symptoms of COVID19 due to SARS-CoV-2 infection

   a. Symptoms Defined as: Fever, Dry cough, Fatigue, Difficulty breathing, Sore throat, Diarrhea, Rhinorrhea (runny nose), or new aches/pains.
2. Ongoing symptoms not due or not known to be due to SARS-CoV-2 infection

   a. Symptoms Defined as: Fever, Dry cough, Fatigue, Difficulty breathing, Sore throat, Diarrhea, Rhinorrhea (runny nose), or new aches/pains.
3. Patients receiving ongoing medical symptomatic treatment or prophylaxis treatment related to COVID-19 due to SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals cared for at Froedtert Hospital, Milwaukee, Wisconsin who meet the inclusion and exclusion criteria as outlined.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Characterization of specific T cell responses in peripheral blood isolated from patients that have been exposed to SARS-CoV-2. | Up to 1 year post infection.